

# **ETOP 7-14 NICHE**

# Afatinib in pretreated patients with advanced NSCLC harbouring HER2 exon 20 mutations

**Sponsor: European Thoracic Oncology Platform (ETOP)** 

# STATISTICAL ANALYSIS PLAN - FINAL ANALYSIS

| SAP VERSION | 2.1 |
|-----------------------------|------------------------------------|
| SAP VERSION DATE | 23 January 2017 |
| TRIAL STATISTICIANS | Urania Dafni, Zoi Tsourti |
| TRIAL PRIMARY INVESTIGATORS | Rafal Dziadziuszko, Solange Peters |
| SAP AUTHOR | Zoi Tsourti |
| APPROVED BY | Urania Dafni |

# **TABLE OF CONTENTS**

| 1. | INT | RODUCTION | 3 |
|----|-------|--------------------------------------------------|-----|
| | 1.1 | Preface | 3 |
| | 1.2 | History of the Study | 3 |
| | 1.3 | Purpose of the present Statistical Analysis Plan | 4 |
| 2. | GEN | NERAL CONSIDERATIONS FOR THE ANALYSIS | 4 |
| | 2.1 | Timing of Analysis | 4 |
| | 2.2 | Analysis Populations | . 4 |
| | 2.3 | Statistical Considerations | 5 |
| | 2.4 | Missing Data | 5 |
| 3. | SUN | MMARY OF STUDY DATA | 5 |
| | 3.1 | MAIN OUTCOME | 5 |
| | 3.2 | Baseline characteristics | . 6 |
| | 3.3 | Follow-up and treatment administration | 6 |
| | 3.4 | Translational results | . 6 |
| 4. | EFF | ICACY ANALYSIS | . 6 |
| 5. | SAF | ETY ANALYSIS | 7 |
| 6. | REP | PORTING CONVENTIONS | 8 |
| 7. | TEC | HNICAL DETAILS | 8 |
| 8. | LIST | TING OF TABLES AND FIGURES | 8 |
| Δ | PPFND | IX | 16 |

#### 1. INTRODUCTION

#### 1.1 Preface

Afatinib presents a manageable toxicity profile and potentially offers a significant activity in terms of disease control and long-term outcome. Therefore this treatment option offers a good benefit to risk ratio in patients with HER2-mutate advanced NSCLC.

The primary objective of the study is to evaluate the ability of afatinib to control disease in pretreated patients with advanced NSCLC harbouring HER2 exon 20 mutations. More particularly, the primary endpoint is disease control at 12 weeks.

The secondary objectives of the study are:

- To evaluate secondary measures of clinical efficacy including progression-free survival (PFS),
- To assess the safety and the tolerability of the treatment.

# 1.2 History of the Study

ETOP/7-14 NICHE trial was activated in December 2014 and the first patient was enrolled on September 2015.

The ETOP IDMC reviewed the trial safety data during its scheduled bi-annually meetings, in April 2016 (n=5 patients enrolled; no safety issues identified) and October 2016 (n=13) when the interim analysis was presented. Follow-up was suspended based on the interim analysis and an unscheduled follow-up IDMC meeting in November 2016 on the 13 enrolled patients enrolled).

At the IDMC meeting of October 2016, the interim analysis (1st stage of Simon's two-stage design) was presented. Among the first 9 patients, 5 patients (55.6%) had not reached week 12 free of progression. Thus, the stopping threshold of the 1st stage of Simon's two-stage design was reached, since more than the maximum allowed of 3 patients had a progression by 12 weeks. Based on these results, the IDMC recommended suspending further recruitment into the trial while continuing the treatment and close follow-up for the enrolled patients.

A follow-up analysis, once all enrolled patients reached the 12-week assessment, was performed in November 2016. Among all 13 enrolled patients, 6 patients (46.2%) had not reached week-12 free of progression.

Based on the data and results of the interim analysis and considering the protocol specified early stopping rule, the IDMC recommended that:

- The ETOP 7-14 NICHE trial should be permanently closed to accrual.
- Treatment and follow-up of enrolled patients may continue based on the judgement of the treating physician.
- Patients should be informed.

# 1.3 Purpose of the present Statistical Analysis Plan

The purpose of the present Statistical Analysis Plan (SAP) is to provide an analytic and solid framework for the final analysis of the patients enrolled in the NICHE study.

More details on the planned final evaluation in terms of methods, reporting conventions and formats are described in detail in the following sections.

The overall objectives and methods of the study, as dictated by its protocol, may be found in the Appendix.

# 2. GENERAL CONSIDERATIONS FOR THE ANALYSIS

# 2.1 Timing of Analysis

The final analysis will be performed at least six months after the last patient was enrolled and as soon as the database is formally locked.

# 2.2 Analysis Populations

# Interim evaluation Cohort

The interim evaluation cohort will include the first 9 patients enrolled in the study, which were used for the evaluation of Simon's stage one.

# Efficacy Cohort

The efficacy cohort will include all eligible patients enrolled in the study until trial termination.

# Safety Cohort

The safety cohort will encompass all eligible enrolled patients who have received at least one dose of trial treatment.

#### 2.3 Statistical Considerations

Primary endpoint is disease control (DC), defined as complete (CR) or partial response (PR), or disease stabilisation (SD) lasting at least 12 weeks.

Simon's two stage phase II design has been adopted. A Disease Control Rate (DCR) of 50% was considered as unacceptable, targeting a DCR of 75%. Hence the null hypothesis under consideration was that the DCR≤50% versus the alternative that DCR≥75%. For a one-sided type I error of 10% and power of 80%, a total of 22 patients were needed, with 9 patients in the first stage. If in the first stage, 6 out of the 9 patients achieved Disease Control, then the trial would proceed to the second stage and recruit an additional 13 patients for a total of 22 patients. If at least 14 out of the 22 patients achieved Disease Control, then this finding would indicate that it would be reasonable to proceed to a Phase III trial.

Secondary endpoints include objective response (OR), defined as best overall response (CR or PR, using RECIST 1.1 criteria) across all assessment time-points during the period from enrolment to termination of trial treatment, progression-free survival (PFS), defined as the time from the date of enrolment until documented progression or death, overall survival (OS), defined as time from the date of enrolment until death from any cause (censoring occurring at the last follow-up date), and toxicity as specified by the adverse events classified according to NCI CTCAE version 4.

# 2.4 Missing Data

Missing values will not be replaced by any statistics calculated over non-missing data.

# 3. SUMMARY OF STUDY DATA

# 3.1 MAIN OUTCOME

The primary endpoint according to study's protocol, is the **DCR**.

DCR will be calculated along with 90% exact binomial confidence interval (CI) for the efficacy cohort.

PFS and OS (medians and rates) will be estimated based on the product-limit Kaplan-Meier method, while the corresponding 95% CIs for the median values will be based on the complementary log-log transformation.

#### 3.2 Baseline characteristics

Baseline characteristics will be summarized and presented overall **for all enrolled patients.** 

All continuous variables will be summarised using the following descriptive statistics: n (non-missing sample size), mean, 95% CI for the mean, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures.

# 3.3 Follow-up and treatment administration

Follow-up time will be defined as time between the minimum of enrolment and start treatment date and last contact date. The median follow-up will be estimated based on reverse censoring of overall survival.

Time-to-Treatment Failure (TTF) will also be calculated based on the Kaplan-Meier method, and the specific reasons of treatment failures will be provided.

#### 3.4 Translational results

The results of all translational analyses (of the tests performed centrally) in the frame of the study we be analytically presented in tabular format.

#### 4. EFFICACY ANALYSIS

The primary efficacy analysis will include all eligible enrolled patients.

The primary endpoint is disease control, defined as complete or partial response or disease stabilisation lasting at least 12 weeks.

Results on the primary endpoint will be presented for the whole efficacy cohort as well as for the 'interim analysis' cohort.

Objective response, progression-free survival and overall survival, the secondary efficacy endpoints of the NICHE trial, will also be evaluated for the whole efficacy cohort.

Best overall response, defined as best response across all assessment time-points, during the period from enrolment to termination of trial treatment, and objective response rate, defined as the best overall response (complete or partial response) will be summarized in table format.

PFS (defined as the time between the minimum of enrolment and start treatment date until documented progression or death) and OS (defined as the time between the minimum of enrolment and start treatment date until death or last contact date for censored patients) will be summarized through tables as well as graphically depicted via Kaplan-Meier curves and alternative graphical illustrations if possible (spider plot, swimmer plot).

As an exploratory analysis, the association of the primary endpoint (Disease control at 12 weeks) with patients' baseline characteristics, prior treatments received as well as with translational results will be also investigated.

More particularly, the distribution of patients' baseline characteristics and prior treatments will be presented separately for the group of patients that achieved disease control at 12th week versus the group of patients that did not achieve disease control and corresponding Fisher's exact tests will be provided.

In a similar manner, all translational results will be presented separately for the groups of patients that achieved or not disease control. Also, PFS and OS results will be provided for selected subgroups of patients with particular interest (type of ERBB2 mutation, Gender and Smoking status). Log-rank test comparing the survival curves between subgroups will be also presented.

# **5. SAFETY ANALYSIS**

The safety cohort will encompass all patients who have received at least one dose of trial treatment. Safety and tolerability of the afatinib treatments will be described by tabulation of the CTCAE V4 grade. In particular, safety analysis will include assessment of the experience of adverse events (AE) and serious adverse events (SAE), the frequency of AEs, the numbers of patients experiencing specific number of adverse events and their distribution by CTCAE V4 grade. Further exploration on AEs, with respect to their grade will include the presentation of maximum severity of AEs for each patient as well as the distribution of worst degree of severity by patient.

Note: If the same adverse event is recorded more than once for a specific patient, it will be counted only once keeping the one with the higher grade.

For a closer investigation and for purposes of medical review, information on AEs will also be provided by patient. This information will consist of AE description and grade, date of AE onset and end date (if the event is resolved), its potential relation to treatment and his/her specific outcome.

A summary table of all the narratives of patients with SAE will also be provided.

Furthermore, the baseline symptoms experienced by some of the patients, which are not counted as adverse events –unless their grade was increased or they appeared as new events at a later period of time- will be presented separately.

# 6. REPORTING CONVENTIONS

P-values≥0.001 will be reported with two significant digits (e.g. p=0.26, p=0.026, p=0.003); p-values less than 0.001 will be reported as "<0.001". The mean, 95% confidence limits, quantiles, and any other statistics, will be reported to one decimal. Hazard ratios (HRs) and their 95% CI's will be reported to two decimals. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 decimals.

# 7. TECHNICAL DETAILS

Data will be analyzed using the SAS software package (version 9.4). The use of R language will also be considered for the production of specific plots.

A second statistician, the **reviewing statistician** will independently reproduce all analysis and summary statistics. The **reviewing statistician** will have an overview of the entire analysis and will explicitly check the code producing tables and figures as well as any other pieces of code as desired.

# 8. LISTING OF TABLES AND FIGURES

Table 1 gives a tabulation of the following aspects unique to each table:

- Title
- Numbering
- Population
- Endpoint(s)

Time Points or details of how to conglomerate multiple observations

- Covariates or Subgroups used to break down summary statistics
- Which summary statistics will be calculated

For figures the equivalent information is summarized in Table 2 and includes the following:

- Title
- Numbering
- Population
- Type of figure
- Endpoint(s), and which is used for horizontal and vertical co-ordinates
- Statistic(s) used in calculating co-ordinate values used in the figure
- Covariates used within the figure used to determine colours or symbols

**Table 1.** Listing of Tables

| Table title | Number | Population | Endpoint | Time Points<br>or how to<br>conglomerate | Covariates or<br>Subgroups | Summary<br>Statistics | Formal<br>Analysis | Notes |
|---|---|---|---|---|---|---|---|---|
| Section I: Patient Accru | al & Baseli | ne Characteri | stics | | | | | |
| Accrual by center | Accrual by center 1 Efficacy cohort | | Accrual | NA | center | n (%) | NA | Sorted by descending "n" |
| Patient and tumor<br>baseline characteristics | atient and tumor 2 Efficacy Smoking histor schort ECOG Performation enrolment) TNM staging | | Smoking history<br>ECOG Performance status (at<br>enrolment) | Baseline | - | n (%) | NA | |
| Information on previous and subsequent lines of treatment | 3 | Efficacy<br>cohort | Type of prior platinum treatment Afatinib Treatment Line Further treatment Type of further treatment | Baseline,<br>Follow-up | - | n (%) | NA | |
| History of previous diseases/conditions | 4 | Efficacy<br>cohort | Types of previous diseases and conditions | Baseline | - | n (%) | NA | |
| Results of HER2 central testing | 5 | Efficacy<br>cohort | HER2 (ERBB2) mutation | Baseline | - | n (%) | NA | |
| Section II: Follow-up & | Treatment | | on | | | ı | 1 | |
| Time on follow-up and Time on treatment 6 | | Efficacy<br>cohort | No. of patients still on f-up, no.<br>of discontinuations | End of follow-<br>up | - | n (%)<br>median, interq.<br>range | Reverse<br>Censoring<br>based on<br>OS (f-up)<br>Kaplan –<br>Meier<br>analysis<br>(both) | |
| Reasons of treatment failures Section III: Analysis of I | 7<br>Primary En | Efficacy<br>cohort<br><b>dpoint</b> | Reasons of treatment failures | | | n (%) | NA | |

| Table title | Number | Population | Endpoint | Time Points<br>or how to<br>conglomerate | Covariates or<br>Subgroups | Summary<br>Statistics | Formal<br>Analysis | Notes |
|---|---|---|---|---|---|---|---|---|
| Disease Control Rate<br>(DCR) at 12 weeks | 8 | Interim evaluation cohort & Efficacy cohort | Disease Control (Yes / No) | 12-week<br>evaluation<br>(tumor<br>assessment) | - | n (%) | NA | |
| Section IV: Analysis of S | | | | | | 1 | | |
| Best Overall Response<br>and Objective Response<br>Rate (ORR) for all<br>enrolled patients<br>(N=13) | 9 | Efficacy<br>cohort | Best Overall Response, ORR | OR: The best overall response (CR or PR) across all assessment time-points according to RECIST Criteria 1.1, during the period from enrolment to termination of trial treatment. | | n (%) | | |
| Progression-free<br>Survival (PFS) for all<br>enrolled patients<br>(N=13) | 10 | Efficacy<br>cohort | PFS | PFS: time from the date of enrolment until documented progression or death without documented progression | - | KM estimates: no. of patients, n(%) of PFS events, 12-week PFS (%) (95% CI), median PFS (in weekw) | Kaplan –<br>Meier<br>analysis | |
| Overall Survival (OS)<br>for all enrolled patients<br>(N=13) | 11 | Efficacy<br>cohort | OS | OS: time from<br>the date of<br>enrolment<br>until death | - | KM estimates:<br>no. of patients,<br>n(%) of deaths,<br>xx-weeks OS | Kaplan –<br>Meier<br>analysis | |

| Table title | Number | Population | Endpoint | Time Points<br>or how to<br>conglomerate | Covariates or<br>Subgroups | Summary<br>Statistics | Formal<br>Analysis | Notes |
|---|---|---|---|---|---|---|---|---|
| | | | | from any<br>cause | | (%) (95% CI),<br>median OS (in<br>weeks) | | |
| Section V: Translationa | | | | | 1 | | | |
| Translational results of central testing | 12 | Efficacy<br>cohort | All biomarkers included in the central testing (wild-type, mutation detected, type of mutation detected) | Baseline | - | n (%) | | |
| Section VI: Exploratory | Analysis of | f Efficacy End <mark>p</mark> | | | | | | |
| Primary endpoint by baseline characteristics | 13 | Efficacy<br>cohort | DC at 12w achieved or not for<br>each value of baseline<br>characteristics | 12-week<br>assessment | Different values<br>of baseline<br>characteristics | n (%) | Fisher's exact test | |
| Primary endpoint by prior treatment | 14 | Efficacy<br>cohort | DC at 12w achieved or not for each value of prior treatment | 12-week<br>assessment | Different types<br>of prior<br>treatment | n (%) | Fisher's exact test | |
| Primary endpoint by translational results | 15 | Efficacy<br>cohort | DC at 12w achieved or not for<br>each value of biomarkers<br>centrally tested | 12-week<br>assessment | Different status<br>of biomarkers<br>tested | n (%) | Fisher's exact test | |
| Progression-free<br>survival (PFS) for<br>selected subgroups of<br>patients | 16 | Efficacy<br>cohort | PFS | PFS: time from the date of enrolment until documented progression or death without documented progression | ERBB2, gender,<br>smoking status | KM estimates: no. of patients, n(%) of PFS events, 12-week PFS (%) (95% CI), median PFS (in weekw) | Kaplan –<br>Meier<br>analysis | |
| Overall survival (OS)<br>for selected subgroups<br>of patients | 17 | Efficacy<br>cohort | OS | OS: time from the date of enrolment until death from any cause | ERBB2, gender,<br>smoking status | KM estimates: no. of patients, n(%) of deaths, xx-weeks OS (%) (95% CI), median OS (in weeks) | Kaplan –<br>Meier<br>analysis | |

| Table title | Number | Population | Endpoint | Time Points<br>or how to<br>conglomerate | Covariates or<br>Subgroups | Summary<br>Statistics | Formal<br>Analysis | Notes |
|---|---|---|---|---|---|---|---|---|
| Section VII: Safety Anal | ysis | | | | | | | |
| (Serious) Adverse<br>event overview | 18 | Safety<br>cohort | AE / SAE | At the end of each treatment visit, Within 24h of occurrence of SAE | - | n (%) of persons who have experienced >=1 AE or SAE | - | |
| Number of patients experiencing specific number of adverse events | 19 | Safety<br>cohort | AE | At the end of each treatment visit | - | n (%) | - | |
| Number of patients<br>experiencing specific<br>number of serious<br>adverse events | 20 | Safety<br>cohort | SAE | At the end of each treatment visit, Within 24h of occurrence of SAE | - | n (%) | - | |
| Maximum severity of adverse events (AE/SAE) per patient | 21 | Safety<br>cohort | AE / SAE | At the end of each treatment visit, Within 24h of occurrence of SAE | - | n (%) | | |
| Distribution of adverse<br>events (AE/SAE) by<br>Grade | 22 | Safety<br>cohort | AE / SAE | At the end of each treatment visit, Within 24h of occurrence of SAE | Severity grade<br>(NCI CTCAE<br>version 4) | n (%) | - | In case of multiple reports of the same AE/SAE (grouped according to CTCAE V4) for a particular patient, the |

| Table title | Number | Population | Endpoint | Time Points<br>or how to<br>conglomerate | Covariates or<br>Subgroups | Summary<br>Statistics | Formal<br>Analysis | Notes |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | | event is counted once. |
| Baseline symptoms by patient | 23 | Safety<br>cohort | AE | At baseline | - | - | - | Patients ordered<br>by enrolment<br>date |
| Adverse event information by patient | 24 | Safety<br>cohort | AE / SAE | At the end of each treatment visit, Within 24h of occurrence of SAE | - | - | - | Patients ordered<br>by enrolment<br>date |
| Narratives of patients with SAE | 25 | Safety<br>cohort | SAE | At the end of each treatment visit, Within 24h of occurrence of SAE | - | - | - | Patients ordered<br>by enrolment<br>date |

 Table 2. Listing of Figures

| Title | Number | Population | Type of graph | Horizontal<br>Variables | Vertical<br>Variables | Groupings | Notes |
|---|---|---|---|---|---|---|---|
| Section I: Patient Accru | al & Baseline | Characteristics | | | | | |
| Expected vs Observed<br>Accrual | 1 | Efficacy cohort | Line graph | time | cumulative<br>number of<br>patients | - | - |
| Section II: Follow-up & | Treatment A | dministration | | | | | |
| Kaplan Meir plot for<br>Time-to-Treatment<br>Failure (TTF) | 2 | Efficacy cohort | KM | time | probability | - | - |
| Section IV: Analysis of S | Secondary Eff | icacy Endpoints | | | | | |
| Plot of tumor response | 3 | patients in efficacy<br>cohort evaluable for<br>tumor-response | Spider plot | time | % change (in<br>sum of<br>diameter of<br>target<br>lesions) from<br>baseline | | It depends on the data<br>whether it will be<br>feasible to produce it |
| Plot of duration of tumor response | 4 | patients in efficacy<br>cohort evaluable for<br>tumor-response | Swimmer<br>plot | Duration of response (in weeks) | Patient id | - | It depends on the data<br>whether it will be<br>feasible to produce it |
| Kaplan Meir plot for<br>Progression Free<br>Survival (PFS) | 5 | Efficacy cohort | KM | time | probability | - | - |
| Plot of Progression-free<br>Survival by patient,<br>according to primary<br>endpoint (disease<br>achieved at 12 weeks) | 6 | Efficacy cohort | Bar-plot | Patient id | PFS (in weeks) | - | Additional patients' characteristics will be shown below the bars |
| Kaplan Meir plot for<br>Overall Survival (OS) | 7 | Efficacy cohort | KM | time | probability | - | - |

# **APPENDIX**

# IMPORTANT INFORMATION AS DESCRIBED IN THE PROTOCOL

#### Objectives

The **primary objective** of the study is to evaluate the ability of afatinib to control disease in pretreated patients with advanced NSCLC harbouring HER2 exon 20 mutations. More particularly, the primary endpoint is **disease control at 12 weeks.** 

# Secondary objectives

The secondary objectives of the study are:

- To evaluate secondary measures of clinical efficacy including progression-free survival (PFS),
- To assess the safety and the tolerability of the treatment.

#### **Endpoints**

- 1. Primary endpoint: Disease control at 12 weeks
- 2. Secondary endpoints:
  - a. Progression-free survival by RECIST v1.1
  - b. Objective response rate by RECIST v1.1
  - c. Overall survival
  - d. Adverse events graded according to CTCAE V4.0

# Most important eligibility criteria

#### Inclusion criteria at enrolment:

- Histologically or cytologically confirmed, non-predominant squamous subtype,
  - Stage IIIB (non amenable to curative-intent multimodal treatment) or IV NSCLC, according to 7th TNM classification
  - Tumour is platinum-refractory
  - Measurable or evaluable disease (according to RECIST 1.1 criteria)
  - Locally documented HER2 mutation
  - Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
  - Life expectancy >3 months
  - Adequate haematological, renal and hepatic function
  - Effective contraception, no pregnancy

#### Exclusion criteria at enrolment:

- Mixed small-cell and non-small-cell histologic features
- Uncontrolled lepto-meningeal metastatic disease
- Previous treatment with HER2 targeted antibody or tyrosine kinase inhibitor
- Any previous (in the past 3 years) or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ ductal carcinoma of the breast
- History or presence of clinically relevant cardiovascular abnormalities

• Other serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical processes that could affect the patient's capacity to participate in the trial

- Interstitial lung disease or pulmonary fibrosis
- Any concurrent systemic anticancer therapy

#### Treatment

Afatinib 40 mg p.o./day until tumour progression or lack of tolerability



SCHEMA 1. Trial design

**Population:** Advanced stage NSCLC, harbouring *HER2* exon 20 mutations.

Design: A Phase II single-arm multicenter trial

Planned sample size: 22 patients

Total trial duration: 40 months from enrolment of the first patient, including 6 months of follow-up from

enrolment of the last patient

# Statistical considerations

Simon's two stage phase II design is adopted. A Disease Control Rate (DCR) of 50% is considered as unacceptable, targeting a DCR of 75%. Hence the null hypothesis under consideration is that the DCR≤50% versus the alternative that DCR≥75%. For a one-sided type I error of 10% and power of 80%, a total of 22 patients are needed, with 9 patients in the first stage. If in the first stage, 6 out of the 9 patients achieve Disease Control, then the trial will proceed to the second stage and recruit an additional 13 patients for a total of 22 patients. If at least 14 out of the 22 patients achieve Disease Control, then this finding will indicate that it would be reasonable to proceed to a Phase III trial.